CLINICAL TRIAL: NCT03030300
Title: Remission Rate of Newly Diagnosed Type 2 Diabetes Outpatients Treated With Short-term Intensive Insulin Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lin Liao, chief of endocrinology department at Qianfoshan Hospital, Qianfoshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: qfsnfm-005
Record Dates: First submitted 2017-01-02; First posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Type2 Diabetes
Keywords: type 2 diabetes; remission; short-term intensive insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Novolin 30R;Pioglitazone;Metformin (Experimental): Drugs: Insulin (Novolin 30R) monotherapy or combined with one or two oral drugs (metformin 0.5 mg tid and pioglitazone hydrochloride 15 mg qd).
  Interventions: Drug: Novolin 30R;Pioglitazone;Metformin

INTERVENTIONS:
Drug: Novolin 30R;Pioglitazone;Metformin — * Insulin (Novolin 30R) was titrated according to the level of blood glucose until reached euglycemia (FPG≤6.1mmol/L and/or P2hBG≤8.0mmol/L and/or HbA1c ≤6.5%). After glucose was well controlled within these targets for 4 weeks, insulin dosage was gradually decreased until discontinued;
  * Pioglitazone hydrochloride was discontinued if the glucose was well controlled at the 6th week after the cessation of insulin;
  * Metformin was the last drug that to be discontinued if the glucose was still well controlled at the 4th week after the cessation of pioglitazone.

SUMMARY:
To evaluate the long-term remission rate of short-term intensive insulin (STII) therapy in newly diagnosed type 2 diabetes outpatients and investigate the predictors contributing to the remission rate.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, insulin-naive type 2 diabetes outpatients
* Diabetes duration less than 1 year

Exclusion Criteria:

* Various acute complications
* Hepatic transaminase >2.5x normal reference value (glutamic-pyruvic transminase>100U/L, glutamic-oxalacetic transaminase > 100U/L)
* Abnormal renal functions (serum cretinine>the normal reference value)
* Cardiac insufficiency (America NYHA caediac function >3)
* Type 1 diabetes mellitus
* Ongoing hormone therapy
* Women in gestation and lactation
* Patients with other endocrine disorders

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2008-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
prolonged-remission rate | 5 years
  hyperglycemia below diagnostic thresholds for diabetes without active pharmacologic therapy or ongoing procedures of 5 years' duration.
partial-remission rate | 5 years
  hyperglycemia below diagnostic thresholds for diabetes without active pharmacologic therapy or ongoing procedures of more than 3 months' duration, and less than 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Liao, MD, Study Chair — Qianfoshan Hospital
Locations (3):
- China (3):
  - Shandong Provincial Hospital, Jinan, Shandong
  - Qianfoshan Hospital, Jinan, Shandong
  - Qilu Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: Undecided